CLINICAL TRIAL: NCT07319377
Title: A Multicenter, Prospective, Randomized, Parallel-Group, Assessor-blinded, Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of a Digital Therapeutic Device for Improving Muscle Strength in Patients With Sarcopenia
Brief Title: Evaluation of Safety and Efficacy of a Digital Therapeutic Device to Improve Strength in Sarcopenia (Sarc-DTx)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Exosystems (Industry)
Collaborators: The Catholic University of Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC25DDDS0072
Record Dates: First submitted 2025-11-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Device Group (Home-based DTx exercise group after training) (Experimental): Participants perform personalized resistance exercises using a digital therapeutic device (mobile application) at home for 12 weeks, with sessions conducted at least 3 times per week, 50 minutes per session (≥150 minutes/week). The program includes exercise automatic intensity adjustment, exercise recording/analysis, and physician monitoring
  Interventions: Device: exoDTx
- Control Group (Self-exercise) (Active Comparator): No mobile application is used. Participants perform the same type of exercise using QR code-based educational materials, self-regulating their exercise time, at least 3 times per week, 50 minutes per session, for a total of 12 weeks, with frequency and duration identical to the experimental group.
  Interventions: Behavioral: Self-exercise (Educational Material)

INTERVENTIONS:
Device: exoDTx — Experimental group (exoDTx): After baseline on-site training, participants perform personalized resistance exercises at home using a mobile app ≥3 times/week, 50 min/session, for 12 weeks (≥150 min/week). The program provides grip strength-based automatic intensity adjustment, exercise recording, feedback, and physician monitoring.
  Delivery: Nonpharmacological, non-invasive, home-based exercise program. The experimental group uses a mobile app; the control group uses educational materials.
  Initial instruction occurs on-site. Visits & Monitoring: Screening/Baseline (week 0), In-treatment (weeks 4, 8), Post-treatment (week 12), and Follow-up (week 24).
  Arms: Experimental Device Group (Home-based DTx exercise group after training)
Behavioral: Self-exercise (Educational Material) — Control group (Self-exercise): No app is used. Participants perform the same exercise guided by QR code-based educational materials, ≥3 times/week, 50min/session, for 12 weeks, maintaining exercise logs without automatic adjustment or remote monitoring.
  Delivery: Non-pharmacological, non-invasive, homebased exercise program. The experimental group uses a mobile app; the control group uses educational materials. Initial instruction occurs on-site. Visits & Monitoring: Screening/Baseline (week 0), In-treatment (weeks 4, 8), Post-treatment (week 12), and Follow-up (week 24).
  Arms: Control Group (Self-exercise)

SUMMARY:
This clinical trial aims to demonstrate that the use of a digital therapeutic device (exoDTx) in patients with sarcopenia is superior to self-exercise in terms of muscle strength improvement and safety.

DETAILED DESCRIPTION:
Background Sarcopenia is a condition characterized by progressive loss of skeletal muscle mass and strength, which is closely associated with functional decline, falls, and increased mortality.Conventional first-line treatment involves resistance training; however, in older adults, low adherence and practical challenges often limit its effectiveness.Recently, digital therapeutics (DTx) have emerged as promising tools by providing personalized exercise programs, automatic adjustment of intensity, and integrated recording and monitoring functions. These features are expected to overcome the limitations of selfdirected exercise.Therefore, this study seeks to validate the effectiveness and safety of DTx in improving muscle strength and physical function through a randomized controlled trial (RCT). Research Hypothesis In patients with sarcopenia, the group using digital therapeutics (DTx) will demonstrate superior outcomes in muscle strength improvement and safety compared to the self-exercise group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcopenia according to both the European Working Group on Sarcopenia in Older People (EWGSOP) and the 2019 Asian Working Group for Sarcopenia (AWGS) criteria
* Evidence of reduced muscle strength, defined as handgrip strength < 28 kg for men or < 18 kg for women, or a five-times sit-to-stand test time > 12 seconds without arm support
* Evidence of reduced muscle mass, defined as a skeletal muscle mass index < 7.0 kg/m² for men or < 5.4 kg/m² for women measured by DXA, or < 7.0 kg/m² for men or < 5.7 kg/m² for women measured by BIA
* Ability to independently perform sit-to-stand movements
* Sufficient physical and cognitive ability to participate in the exercise program
* Ability to provide written informed consent
* Ability to operate a mobile phone independently or with assistance from a caregiver

Exclusion Criteria:

* Cognitive impairment defined as a Mini-Mental State Examination score < 20 or inability to participate due to cognitive decline
* Presence of an implanted cardiac pacemaker
* Uncontrolled cardiovascular disease despite appropriate medical treatment
* Lower limb surgery within the past 6 months resulting in inability to walk independently
* Moderate to severe musculoskeletal pain or functional limitations that interfere with objective functional assessments
* Severe obesity defined as a body mass index > 50 kg/m²
* Active cancer treatment or severe systemic frailty
* Hemiplegia resulting in inability to perform the prescribed exercise program
* Anticipated inability to complete the study protocol as determined by the investigator
* Inability to comply with study instructions delivered in Korean

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Change in peak knee extension strength (Nm) from baseline to 12 weeks | 12 weeks after Visit 1 (treatment initiation)
  Between-group comparison of mean change in knee extensor strength measured by lower extremity dynamometer.

SECONDARY OUTCOMES:
Change in peak isometric knee extension strength (Nm) from baseline to 4, 8, and 24 weeks | Baseline, 4 weeks, 8 weeks, and 24 weeks after Visit 1 (treatment initiation)
  To evaluate longitudinal changes in knee extensor muscle strength at weeks 4, 8, and 24 compared with baseline using an lower extremity dynamometer.
Change in body composition (skeletal muscle mass index, fat mass) | 12 weeks after Visit 1 (treatment initiation)
  To evaluate changes in muscle and fat mass measured by bioelectrical impedance analysis (BIA) after 12 weeks of intervention.
Change in Manual Muscle Test (MMT) scores of major limb muscles | 12 weeks after Visit 1 (treatment initiation)
  To assess changes in muscle strength based on standardized MMT grading (0-5 scale) after 12 weeks of intervention..
Change in Fugl-Meyer Assessment (upper/lower extremities; CNS-related sarcopenia subgroup) | 12 weeks after Visit 1 (treatment initiation)
  To examine motor recovery and coordination improvements using the Fugl-Meyer Assessment in participants with CNS-related sarcopenia.
Change in Functional Ambulation Category (FAC) score | 12 weeks after Visit 1 (treatment initiation)
  To assess improvement in walking independence level using the Functional Ambulation Category (0-5 scale).
Change in Berg Balance Scale (BBS) and Timed Up and Go (TUG) performance | 12 weeks after Visit 1 (treatment initiation)
  To evaluate dynamic and static balance performance using BBS score and TUG test time.
Change in Short Physical Performance Battery (SPPB) total score and subscores (chair stand, gait speed, balance) | 12 weeks after Visit 1 (treatment initiation)
  To assess lower extremity function using SPPB, including 5-time chair stand, 6-meter gait speed, and balance tests.
  SPPB - 5-time chair stand (time) 6-meter gait speed (SPPB gait speed) SPPB balance - score SPPB balance - time in seconds
Change in Muscle Function Index (MFI) from surface EMG analysis | 12 weeks after Visit 1 (treatment initiation)
  To quantify changes in muscle fatigue characteristics derived from surface electromyography (EMG) during resistance exercises.
Change in Strength, Assistance with walking, Rise from a chair, Climb stairs, and Falls (SARC-F) Questionnaire Score | Baseline, 4 weeks, 8 weeks, 12 weeks, and 24 weeks
  To assess changes in self-reported sarcopenia risk using the full Strength, Assistance with walking, Rise from a chair, Climb stairs, and Falls (SARC-F) questionnaire. The SARC-F consists of 5 items, each scored from 0 to 2, resulting in a total score ranging from 0 to 10, with higher scores indicating worse sarcopenia severity and greater functional limitation.
Change in Sarcopenia Quality of Life (SarQOL) score | Baseline, 4 weeks, 8 weeks, 12 weeks, and 24 weeks
  To measure sarcopenia-specific quality of life changes using SarQOL total score and domain subscores.
  SarQOL contains 55 items generating a total score from 0 to 100, with higher scores indicating better quality of life.
Change in Self-Efficacy for Home Exercise Programs Scale score | 12 weeks after Visit 1 (treatment initiation)
  To evaluate participants' confidence in independently performing prescribed home-based exercises.
System Usability Scale (SUS) total score of the exoDTx mobile application | 12 weeks after Visit 1 (treatment initiation)
  To assess user satisfaction and perceived usability of the exoDTx digital therapeutic application using SUS.

CONTACTS AND LOCATIONS:
Overall Officials: Sangui Choi, CPO, Principal Investigator — Exosystems
Locations (3):
- South Korea (3):
  - Bucheon St. Mary's Hospital, Bucheon-si
  - Seoul St. Mary's Hospital, Seoul
  - St.Vincent's hospital, Suwon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Song K, Eun Shin H, Park W, Lee D, Jang J, Yang Shim G, Choi S, Kim M, Lee H, Won Won C. Digital Biomarker for Muscle Function Assessment Using Surface Electromyography With Electrical Stimulation and a Non-Invasive Wearable Device. IEEE Trans Neural Syst Rehabil Eng. 2024;32:3048-3058. doi: 10.1109/TNSRE.2024.3444890. Epub 2024 Aug 26. PMID 39150814